CLINICAL TRIAL: NCT05646238
Title: The Effect of Psychoeducation Based on Leventhal's Self-Regulation Model on Dysmenorrhea in Nursing Students: A Single-Blind Randomized Controlled Study
Brief Title: The Effect of Psychoeducation on Dysmenorrhea in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Merve Işık, research assistant doctor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gaziuni.
Record Dates: First submitted 2022-11-30; First posted 2022-12-12 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Dysmenorrhea
Keywords: coping; nursing care; student; psychoeducation; dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental design
Who Masked: Participant
Masking Description: Those with a VAS score of 4 and above were assigned to the experimental and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Students assigned to the experimental group will be divided into groups of 6-9. 3 psychoeducation sessions will be held with each group once a week for a total of 3 weeks. Group sessions are estimated to last between 60-75 minutes. Psychoeducational content based on Leventhal's Self-Regulation Model was prepared. In the first stage, cognitive bases of dysmenorrhea, in the second stage, strategies to cope with dysmenorrhea, and in the third stage, the effectiveness of coping strategies in dysmenorrhea will be discussed. In the second stage, the participants will be taught the progressive muscle relaxation exercise, which is among the strategies to cope with dysmenorrhea. Sessions will be held online.
  Interventions: Other: psychoeducation
- control group (Active Comparator): The control group will be given a online training of 30-45 minutes covering dysmenorrhea and coping in a single session. From the first menstrual cycle after the training session is completed, measurements will be made in 3 consecutive menstrual cycles.
  Interventions: Other: training

INTERVENTIONS:
Other: psychoeducation — Students assigned to the experimental group will be divided into groups of 6-9. 3 psychoeducation sessions will be held with each group once a week for a total of 3 weeks. Group sessions are estimated to last between 60-75 minutes. Psychoeducational content based on Leventhal's Self-Regulation Model was prepared. In the first stage, cognitive bases of dysmenorrhea, in the second stage, strategies to cope with dysmenorrhea, and in the third stage, the effectiveness of coping strategies in dysmenorrhea will be discussed. In the second stage, the participants will be taught the progressive muscle relaxation exercise, which is among the strategies to cope with dysmenorrhea. Sessions will be held online.
  Arms: intervention group
Other: training — The control group will be given a online training of 30-45 minutes covering dysmenorrhea and coping in a single session. From the first menstrual cycle after the training session is completed, measurements will be made in 3 consecutive menstrual cycles
  Arms: control group

SUMMARY:
This study will be conducted to examine the effect of psychoeducation based on Leventhal's Self-Regulation Model on dysmenorrhea in nursing students.

DETAILED DESCRIPTION:
This study will be conducted to examine the effect of psychoeducation based on Leventhal's Self-Regulation Model on dysmenorrhea in nursing students.

Hypotheses of the Research

H0a: There is no difference in menstrual pain severity between the experimental group and the control group receiving psychoeducation based on Leventhal's Self-Regulation Model.

H0b: There is no difference between the Functional and Emotional Dysmenorrhea Scale mean scores between the experimental group and the control group receiving psychoeducation based on Leventhal's Self-Regulation Model.

H0c: There is no difference between the Menstruation Symptom Scale mean scores between the experimental group receiving psychoeducation based on Leventhal's Self-Regulation Model and the control group.

Menstrual pain severity in women in the experimental and control groups is the primary result of the study.

Functional and Emotional Dysmenorrhea Scale and Menstruation Symptom Scale mean scores of the women in the experimental and control groups constitute the secondary results of the study.

Type of research The research is a single-center parallel group single-blind randomized controlled experimental study. The study will be conducted in accordance with the CONSORT checklist.

Participants and setting The population of the research will be female students studying at the Nursing Department of Bitlis Eren University. In order to determine the sample size of the study, a power analysis (G*Power 3.1.9.4 version) was conducted by taking the study results of Yılmaz and Şahin (2020), which is similar to our study, as reference. According to the power analysis, the sample size was determined as 62 women in total (d=0.75; α= 0.05; 1-β=90%). However, by calculating the drop out rate (~5%) in the study of Yılmaz and Şahin (2020), 33 women will be included in each group in our study.

Validity-Reliability of the Research Selection bias Inclusion criteria were determined to avoid selection bias. All women who met the following criteria were invited to participate in the study.

Inclusion criteria,

* Having a regular menstrual cycle of 6 months
* Being Nulliparous
* Getting 4 or more points from VAS
* Having smart phone and internet facility
* Having the technical means to use the ZOOM application
* Volunteering to participate in the research Exclusion criteria,
* Having a diagnosis of any gynecological disease
* Having a history of gynecological surgery
* Having an active vaginal infection
* Not having received psychosocial counseling for dysmenorrhea before

Distribution bias (randomization): Simple randomization method will be used in the randomization of the research sample. Participants who are determined to meet the research criteria will be assigned to the experimental and control groups according to the assignment list created through the computer program.

Implementation bias: In this study on implementation bias, participant blinding will be done. For this purpose, an active control group will be used in the research. However, since the implementation of the research will be done by the researchers, the researcher cannot be blinded.

Detection bias (detection bias; How the results were collected): Measures to prevent detection bias will be made using an online questionnaire.

Reporting bias (blinding the person who wrote the report and analyzed the data): The data obtained from the research aimed at preventing reporting bias will be coded as A and B by an independent statistician and transferred to the SPSS program. Analysis of the data will also be done by an independent statistician.

Attrition bias (reduction bias): In case of a decrease in the sample, ITT analysis will be performed.

Data Collection Inclusion Criteria Form, Descriptive Information Form, Visual Analog Scale, Functional and Emotional Dysmenorrhea (Painful Menstruation) Scale and Menstruation Symptom Scale will be used to collect data.

Introductory Information Form; The Introductory Information Form is a 14-question form prepared by the researchers to determine the sociodemographic characteristics (age, income level, family type, longest living place) and characteristics of menstruation and dysmenorrhea (age of menarche, duration of pain, need for analgesic use, analgesics used, applications for pain relief) of the participants.

Visual Analog Scale (VAS); VAS is a one-dimensional scale that is widely used today to measure subjective parameters such as pain intensity. The VAS is a 10 cm long ruler drawn horizontally or vertically, starting with "No pain" and ending with "Unbearable pain". The patient is instructed to place a mark on this line, which corresponds to the severity of the pain, to cross this line. The numerical index of the patient's pain intensity in cm or mm is obtained by measuring the distance from the lowest VAS level to the patient's mark with a ruler. In the VAS, the severity of pain is graded between 0 and 10 points. Usually, "no pain" is rated as 0 points and "worst pain imaginable" is 10 points. Ranges for pain intensity; <3 mild pain, 3-6 moderate pain, >6 severe pain.

Functional and Emotional Dysmenorrhea (Painful Menstruation) Scale; The Functional and Emotional Dysmenorrhea Scale (FEDS) is a Likert-type scale used to evaluate dysmenorrhea functionally and emotionally. Li et al. (2012) Turkish validity and reliability study of the scale was carried out by Gün (2014). The Cronbach's Alpha coefficient of FEDS, which consists of 14 items and two sub-dimensions, is 0.91. Each item is scored between 1 (one) and 5 (five). There is no reverse item in the scale. As the scores obtained from the scale increase, the level of functional and emotional impact of dysmenorrhea also increases.

Menstruation Symptom Scale (MSS); It is a scale developed by Chesney and Tasto in 1975 to evaluate menstrual pain and symptoms. In 2009, Negriff et al. factor structure and usability on adolescents were re-evaluated and updated. Guvenc et al. Turkish validity and reliability were made in 2014 by Güvenç, Seven, & Akyüz, 2014. MSS is a five-point Likert-type scale consisting of twenty-two items. Participants are asked to give a number between 1 (never) and 5 (always) for the symptoms they experience about menstruation. The scale has three sub-dimensions: 'Negative Effects/Somatic Complaints' (Items 1-13), 'Menstrual Pain Symptoms' (Items 14-19) and 'Coping Methods' (Items 20-22). The highest score that can be obtained from the scale is 110, and the lowest score is 22. The MSS score is calculated by taking the total mean score of the items in the scale. An increase in the mean score indicates an increase in the severity of menstrual symptoms. The score obtained from the sub-dimensions is calculated by taking the total score average of the items in the sub-dimensions. The increase in the mean score for the sub-dimensions indicates that the severity of menstrual symptoms related to that sub-dimension increases. The Cronbach's Alpha value of the original scale is 0.86.

Application of Research There will be two groups in the research, namely the experimental and control group. The eligibility of the participants to be included in the study will be determined by using the inclusion criteria form. Introductory Information Form, VAS, Functional and Emotional Dysmenorrhea Scale and Menstruation Symptom Scale will be applied to the participants who are determined to be eligible for inclusion in the study. After filling out the forms, assignments to the groups will be made by randomization.

Experimental group-Intervention group Based on Leventhal's Self-Regulation Model Students assigned to the experimental group will be divided into groups of 6-9. 3 psychoeducation sessions will be held with each group once a week for a total of 3 weeks. Group sessions are estimated to last between 60-75 minutes. Psychoeducational content based on Leventhal's Self-Regulation Model was prepared. In the first stage, cognitive bases of dysmenorrhea, in the second stage, strategies to cope with dysmenorrhea, and in the third stage, the effectiveness of coping strategies in dysmenorrhea will be discussed. In the second stage, the participants will be taught the progressive muscle relaxation exercise, which is among the strategies to cope with dysmenorrhea. Sessions will be held online.

After the completion of the psychoeducation session, measurements will be made in 3 consecutive menstrual cycles, starting from the first menstrual cycle. Measurements will be made on the first day of each menstrual cycle using the VAS, the Functional and Emotional Dysmenorrhea Scale, and the Menstruation Symptom Scale.

Control Group The control group will be given a online training of 30-45 minutes covering dysmenorrhea and coping in a single session. From the first menstrual cycle after the training session is completed, measurements will be made in 3 consecutive menstrual cycles. Measurements will be made on the first day of each menstrual cycle using the VAS, the Functional and Emotional Dysmenorrhea Scale, and the Menstruation Symptom Scale.

ELIGIBILITY:
Inclusion Criteria:

* Having a regular menstrual cycle of 6 months
* Being Nulliparous
* Getting 4 or more points from VAS
* Having smart phone and internet facility
* Having the technical means to use the ZOOM application
* Volunteering to participate in the research

Exclusion Criteria:

* Having a diagnosis of any gynecological disease
* Having a history of gynecological surgery
* Having an active vaginal infection
* Not having received psychosocial counseling for dysmenorrhea before

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female students with dysmenorrhea
Enrollment: 61 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Menstrual pain severity using the Visual Analog Scale | Change from before implementation, 3th week of the practice, at the beginning of menstruation (for 3 months)
  Ranges for pain intensity; <3 mild pain, 3-6 moderate pain, >6 severe pain

SECONDARY OUTCOMES:
Functional and Emotional Dysmenorrhea Scale | Change from before implementation, 3th week of the practice, at the beginning of menstruation (for 3 months)
  There is no reverse item in the scale. Each item is scored between 1 (one) and 5 (five). As the scores obtained from the scale increase, the level of functional and emotional impact of dysmenorrhea also increases.
Menstrual pain severity using the Menstruation Symptom Scale | Change from before implementation and 3th week of the practice, at the beginning of menstruation (for 3 months)
  Scores ranging from 22 to 110 points are obtained in the scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Turkey, Ankara
  - Gazi University, Ankara

REFERENCES:
- [Result] From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO); Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Shazam Hussain M, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke. Int J Stroke. 2018 Aug;13(6):612-632. doi: 10.1177/1747493018778713. Epub 2018 May 22. No abstract available. PMID 29786478
- See also: http://doi.org/10.1016/j.ctim.2019.04.007 — http://doi.org/10.1016/j.ctim.2019.04.007
- See also: http://doi.org/10.1016/j.ejogrb.2010.04.015 — http://doi.org/10.1016/j.ejogrb.2010.04.015
- See also: http://doi.org/10.1016/j.jadohealth.2008.07.018 — http://doi.org/10.1016/j.jadohealth.2008.07.018